CLINICAL TRIAL: NCT02386540
Title: Health Coach Program to Improve Chronic Disease Outcomes Following an Emergency Department Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alameda County Medical Center (Other)
Collaborators: University of California, Berkeley (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Harrison J. Alter, Associate Chair for Research, Department of Emergency Medicine, Highland Hospital, Alameda County Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 14-08123E
Record Dates: First submitted 2015-02-14; First posted 2015-03-12 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Community Health Workers; Community Health Workers: utilization; Emergency Service; Primary Health Care/utilization; Health Services Accessibility
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Health Coaching (Experimental): Patients randomized to the experimental arm receive six months of post-ED health coaching from the Alameda County Health Coach Program (ACHCP) in addition to usual care in the emergency department at enrollment.
  Interventions: Behavioral: Health Coaching
- Usual Care (No Intervention): Patients randomized to the control arm receive usual care in the emergency department at enrollment.

INTERVENTIONS:
Behavioral: Health Coaching — The Alameda County Health Coach program pairs patients with a language-concordant health coach for six months following an ED visit. Health coaches are young adults from the local community employed through Alameda County and trained for three months in topics such as self-management support and motivational interviewing. Health coaches work one-on-one with participants in order to develop an action plan in order to achieve patient-identified health goals. Communication between the health coach and participant includes text messages (weekly), phone calls (twice a month), face-to-face visits (at least once), and accompaniment to a primary care visit (at least once). Health coaches may also assist participants in accessing community resources as related to the individualized action plan.
  Arms: Health Coaching

SUMMARY:
The purpose of this study is to determine whether health coaching initiated in the emergency department (ED) reduces subsequent ED visits, increases primary care visits, and positively impacts health outcomes in patients with diabetes and/or hypertension.

DETAILED DESCRIPTION:
Patients will be recruited by health coaches from the Highland Hospital Emergency Department. Eligible patients who agree to participate will be randomized to the control and experimental groups in a 2:1 ratio respectively because experimental group size is limited by health coach availability and greater loss-to-follow up is expected among the control group. Repeated measures analysis will be used to compare each outcome over the study period. In addition, subgroup analyses will be performed in order to stratify by baseline survey measures or amount of ED visits in the pre-observation period.

ELIGIBILITY:
Inclusion Criteria:

* Willing to work with a health coach
* Plans to reside in Alameda County for the next year
* Has a reliable phone number
* Speaks English or Spanish
* 18 years of age or older
* Meets at least one of the following three criteria: (1) Low medication adherence defined as a continuous medication gap of at least 1 month in the past year OR a new diagnosis of diabetes and/or hypertension; (2) No patient-identified primary care provider (PCP) or no visit to PCP in 1 year; (3) One or more visits to the ED in the last 6 months.

Exclusion Criteria:

* Life-expectancy less than 1 year
* Poorly controlled psychiatric illness
* Homeless
* Active and frequent use of illicit substances
* Currently incarcerated
* Already enrolled in a program for patients with high rates of hospitalization and/or emergency department visits
* Unable to consent due to an unstable condition or serious emotional or neurologic condition
* Admitted or anticipated to be admitted to the hospital from the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Number of emergency department visits | 6 month period after enrollment
  Self-reported measure collected via follow-up phone surveys at 1, 3, and 6 months.

SECONDARY OUTCOMES:
Number of primary care visits | 6 month period after enrollment
  Self-reported measure collected by follow-up phone surveys at 1,3, and 6 months.
Physical health and mental health (Validated measure - SF-12v2) | Baseline, 1 month, 3 months, and 6 months after enrollment
  Validated measure (SF-12v2) collected at baseline and follow-up phone surveys.
Medication adherence (Validated measure - Morisky Medication Adherence Scale, MMAS-8) | Baseline, 1 month, 3 months, and 6 months after enrollment
  Validated measure (Morisky Medication Adherence Scale, MMAS-8) collected at baseline and follow-up phone surveys.
Patient activation (Validated measure - Patient Activation Measure, PAM) | Baseline, 1 month, 3 months, and 6 months after enrollment
  Validated measure (Patient Activation Measure, PAM) collected at baseline and follow-up phone surveys.
Type and frequency of health coach contact | 6 months after enrollment
  Health coach documentation notes will be analyzed to determine the average percent of each type of contact (text, phone, or in-person) and frequency of contact.
Percent of action plan goals achieved (Health coach documentation notes) | 6 months after enrollment
  Health coach documentation notes will be analyzed to determine the percent of goals achieved during the intervention.
Qualitative analysis of action plans (Health coach documentation notes will be analyzed, data will be coded to identify themes such as type of goals, barriers to care, and resources identified in the action plan) | 6 months after enrollment
  Health coach documentation notes will be analyzed using a grounded theory approach, where transcribed data will be coded to identify themes such as type of goals, barriers to care, and resources identified in the action plan.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Freeman-Garrick, MD, Principal Investigator — Highland Hospital - Alameda Health System; Berenice Perez, MD, Principal Investigator — Highland Hospital - Alameda Health System; Harrison Alter, MD, Principal Investigator — Highland Hospital - Alameda Health System
Locations (1):
- Highland Hospital - Alameda Health System, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided